CLINICAL TRIAL: NCT06369090
Title: Effect of Women Breast Size on Lung Monitoring Using Electrical Impedance Tomography
Brief Title: Effect of Breast Size on the Electrical Impedance Tomography Measurement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: JP/1/2013
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Effect of Breast Tissue on EIT Lung Monitoring
Keywords: Breast tissue; Electrical impedance tomography; Regional ventilation

STUDY DESIGN:
Intervention Model Description: Monitoring of 22 subjects, each subject was measured twice with electrode belt in two different positions.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy female volunteers (Experimental): Data were obtained at two phases at supine horizontal position during spontaneous and forced breathing of the volunteers. First, with electrode belt placed over the breast tissue and second, with the electrode belt under the breast tissue.
  Interventions: Device: Electrical impedance tomography (EIT)

INTERVENTIONS:
Device: Electrical impedance tomography (EIT) — Non-invasive, radiation-free bedside lung monitoring using small alternating currents with no known side effects.

SUMMARY:
Twenty-two healthy female volunteers were monitored using electrical impedance tomogprahy (EIT) in two different situations. First, with electrode belt placed over the breast tissue and second, with the electrode belt under the breast tissue. The EIT measurement was performed with adjunct spirometric measurement. The changes of regional ventilation related to the breast tissue and the size of breast tissue were evaluated.

DETAILED DESCRIPTION:
The EIT measurement (PulmoVista 500, Dräger Medical, Germany) was performed in supine lying position. On every subject, an electrode belt of proper size based on the measured thorax circumference was placed. It was crucial to find a right position where it was possible to place the electrode belt over the breast tissue and then underneath the breast tissue, without changing the level and the position of the electrode belt on the thorax. Also, the position of the belt had to be between 4th and 6th intercostal space, as recommended by the manufacturer. The change of the position of the belt relative to the breast tissue was performed in a lying position by a slight pull of the buckled belt away from the subject´s body, so the subject could relocate the breast tissue over the belt using her own hands into the position as desired by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* healthy female volunteers

Exclusion Criteria:

* morbid obesity
* standard exclusion criteria for electrical impedance tomography according to the manufacturer

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The eligibility is based on natural physical differences of the female anatomy.
Enrollment: 22 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2014-05-31 (Actual); Study Completion 2014-05-31 (Actual)

PRIMARY OUTCOMES:
Regional ventilation changes possibly caused by the breast tissue | 30 minutes
  The dependence of the regional ventilation evaluated by EIT on the breast size on the regional ventilation was not confirmed.

SECONDARY OUTCOMES:
Female subjects enrollment in EIT studies and clinical applications | 30 minutes
  Recommendation to include women in studies and clinical applications that use electrical impedance tomography for lung monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Karel Roubik, Prof. Ph.D., Study Director — Faculty of Biomedical Engineering, Czech Technical University in Prague
Locations (1):
- Faculty of Biomedical Engineering, Czech Technical University in Prague, Kladno, Czechia

IPD SHARING:
Plan to Share IPD: No